CLINICAL TRIAL: NCT00840359
Title: Phase 2 Study of the Efficacy of Daylight Activated Photodynamic Therapy in the Treatment of Cutaneous Leishmaniasis
Brief Title: Study of the Efficacy of Daylight Activated Photodynamic Therapy in the Treatment of Cutaneous Leishmaniasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Claes D. Enk, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LeishDAPDT-HMO-CTIL
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; Photodynamic therapy
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Photochemotherapy; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 PDT (Experimental): Leishmania lesion
  Interventions: Procedure: Photodynamic therapy
- Cryo (Active Comparator): Leishmania lesion
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Application of Metvix 16% cream followed by exposure to daylight for 2.5 hours
  Arms: 1 PDT
Procedure: Cryotherapy — Cryotherapy for 2 times 20 sec
  Arms: Cryo

SUMMARY:
The aim of the project is to determine whether daylight activated photodynamic therapy is effective in treating cutaneous leishmaniasis caused by L. major and L. tropical.

PDT is classically performed as a two-step procedure in which MAL application to the lesion constitutes the first step, and PpIX activation by light of appropriate wavelength from an artificial light source constitutes the second step. Based on the knowledge that red and blue light required to activate PpIX are part of the daylight spectrum, the investigators postulated that effective PpIX activation can be obtained by exposure of the MAL treated lesions to daylight thus substantially simplifying the PDT procedure by omitting the 3 hour incubation period and the subsequent exposure to artificial light. In accord, in a recent study the investigators showed that daylight-activated PDT (DA-PDT) was as effective as conventional MAL-PDT in treating precancerous actinic keratoses lesion. Furthermore the investigators found that DA-PDT is significantly less painful than conventional MAL-PDT.

The investigators now propose to study the efficacy of DA-PDT in the treatment of cutaneous leishmaniasis. DA-PDT has obvious advantages to conventional leishmania treatment forms:

As opposed to most of the available treatment options, DA-PDT is a self-administered procedure that does not require the assistance of medical personnel. Secondly, judged by our experience with MAL-PDT, only few treatment sessions are required for effective parasite killing as opposed to the prolonged procedures usually required for treatment of leishmaniasis. Third, PDT has the far the best safety profile of all available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 skin lesions with leishmania caused by L. major or L. tropica

Exclusion Criteria:

* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Eradiation of amastigotes | 3 months following last treatment session

SECONDARY OUTCOMES:
Clinical healing | 3 months following last treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Claes D Enk, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel